CLINICAL TRIAL: NCT00783211
Title: A Placebo Controlled Study of the Efficacy and Safety of Desloratadine vs. Fexofenadine 180 mg. in the Treatment of Subjects With Symptomatic Seasonal Allergic Rhinitis (SAR)
Brief Title: Efficacy and Safety of Desloratadine vs. Fexofenadine 180 mg. vs. Placebo for Treating Seasonal Allergic Rhinitis (SAR)(Study P04053)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P04053
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — desloratadine; fexofenadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): desloratadine
  Interventions: Drug: desloratadine
- 2 (Active Comparator): fexofenadine
  Interventions: Drug: fexofenadine
- 3 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: desloratadine — desloratadine, 5 mg oral tablets, once daily for 15 days
  Other Names: SCH 34117; Clarinex
  Arms: 1
Drug: fexofenadine — fexofenadine, 180 mg tablets, once daily for 15 days; for purposes of blinding, fexofenadine tablets were over encapsulated
  Other Names: Allegra
  Arms: 2
Drug: placebo — placebo, once daily for 15 days
  Arms: 3

SUMMARY:
This was a randomized, double-blind, parallel-group, multicenter study that used both an active control (fexofenadine) and a placebo control to evaluate desloratadine 5 mg once daily during a 15-day treatment period. The active treatments and placebo were allocated in a 2:2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* have demonstrated their willingness to participate in the study and comply with its procedures, including adherence to dosing and visit schedules by signing a written informed consent (the parent/guardian of a subject under 18 years of age also had to sign the informed consent form);
* have been 12 years of age or older, of either sex and any race;
* have had at least a 2-year history (self-reported history was acceptable) of seasonal allergic rhinitis occurring during the same season(s) as the current study;
* have been skin test positive (skin prick test with a wheal diameter at least 3 mm larger than the diluent control or intradermal testing with a wheal diameter at least 7 mm larger than the diluent control) at Screening, or within 12 months prior to the Screening Visit, to an appropriate seasonal allergen, which could include seasonal molds, prevalent in the geographical area of the study site during the study period;
* if female and of childbearing potential (including women who were less than 1 year postmenopausal and women who became sexually active during the study), have been using an acceptable method of birth control (eg, hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (eg, hysterectomy or tubal ligation);
* if female and of childbearing potential, have had a negative urine pregnancy test at Baseline;
* have been free of any clinically significant disease (other than SAR) that would interfere with study evaluations;
* have understood and been able to adhere to the dosing and visit schedules, and agreed to record symptom severity scores, medication times, concomitant medications, and adverse events accurately and consistently in a daily diary;
* have met the following at the Screening Visit: total symptom score (TSS) of 6 or greater (not including congestion), with 2 or more symptoms rated as moderate (2) or severe (3) and no symptom rated as very severe (4) during the 12 hours prior to this visit;
* have met the following on the morning of the Baseline Visit: symptom severity score 7 AM instantaneous TSS of 6 or more (not including congestion), with 2 or more symptoms rated as moderate (2) or severe (3), and no symptom rated as very severe (4).

Exclusion Criteria:

* if female, were pregnant, intended to become pregnant during the study, or were nursing;
* had not observed the designated washout periods for any of the prohibited medications;
* had current evidence of clinically significant hematopoietic, cardiovascular, hepatic, immunologic, renal, neurologic, psychiatric, autoimmune disease, or other disease that precluded the subject's participation in the study; particular attention was to be given to conditions that would interfere with the absorption, distribution, metabolism or excretion of the study drug, or with the subject's ability to complete the diary cards;
* had any clinically significant deviation from normal in the physical examination that, in the investigator's judgment, may have interfered with the study evaluation or affected subject safety;
* were in a situation or condition that, in the opinion of the investigator, may have interfered with optimal participation in the study;
* were participating in any other clinical study(ies);
* were part of the investigational study staff or a family member of the staff personnel directly involved with this study;
* had asthma, with the exception of mild intermittent asthma, ie, controlled with the use of short acting, beta2-agonist adrenoreceptor rescue medication;
* had a current or past history of frequent (2 or more episodes per year for the past 2 years), clinically significant sinusitis or chronic purulent postnasal drip;
* had rhinitis medicamentosa;
* had a history of intranasal drug abuse;
* had a history of hypersensitivity to the study drugs or their excipients, or to Claritin;
* had an upper respiratory tract or sinus infection that required antibiotic therapy with the last dose within 14 days prior to Screening, or had a viral upper respiratory infection within 7 days prior to Screening, or had persistent symptoms at the time of the Screening Visit;
* had nasal structural abnormalities, including nasal polyps easily visible on physical examination and marked septum deviation that significantly interfered with nasal airflow;
* in the opinion of the investigator, were dependent upon nasal, oral or ocular decongestants, nasal topical antihistamines, or nasal steroids;
* if on immunotherapy (desensitization therapy) should not have had a change in dose during the study, and should have remained on the same dose throughout the trial; were not to have received desensitization treatment within 24 hours prior to a visit;
* had been previously randomized into the study at any study site;
* ability to provide informed consent was compromised;
* had a history of non-compliance with medications or treatment protocols;
* had a history of difficulty swallowing pills or had known upper gastrointestinal narrowing or abnormal esophageal peristalsis;
* was a night-shift worker or did not have a standard asleep at night / awake during the day cycle;
* planned to travel outside of the study area during the time of their participation in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2004-08-01 (Actual); Primary Completion 2004-10-01 (Actual); Study Completion 2004-10-01 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of the study treatments with respect to the change from Baseline in the mean AM self-rated instantaneous total symptom score (TSS) (not including nasal congestion) averaged over the 15 days of treatment | 15 days

SECONDARY OUTCOMES:
Change from Baseline in the mean AM/PM self-rated 12-hour reflective TSS (not including nasal congestion) averaged over the 15 days of treatment. | 15 days
Change from Baseline in the mean AM self-rated instantaneous individual symptom scores, including nasal congestion, averaged over the 15 days of treatment. | 15 days
Change from Baseline in the mean AM/PM self-rated 12-hour reflective individual symptom scores, including nasal congestion, averaged over the 15 days of treatment. | 15 days
Joint physician-patient evaluation of response to therapy. | Day 8 and Day 15